CLINICAL TRIAL: NCT00606580
Title: A Pivotal, Randomized, Double-blind, Vehicle-controlled Study to Evaluate WR 279,396 and Paromomycin Alone to Treat Cutaneous Leishmaniasis (in Tunisia)
Brief Title: Phase 3 Study to Evaluate WR 279,396 vs. Paromomycin Alone to Treat Cutaneous Leishmaniasis (in Tunisia)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-14134
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Cutaneous Leishmaniasis
Keywords: cutaneous leishmaniasis, topical treatment, Tunisia
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- WR 279,396 Topical Treament (Experimental): WR 279,396 topical cream (15% paromomycin + 0.5% gentamicin topical cream)
  Interventions: Drug: WR 279,396 topical cream
- Paromomycin Alone Topical treatment (Experimental): Paromomycin Alone topical cream (15% paromomycin topical cream)
  Interventions: Drug: Paromomycin Alone topical cream
- Vehicle Placebo Cream (Placebo Comparator): The cream base without the addition of paromomycin or gentamicin
  Interventions: Drug: Vehicle placebo cream

INTERVENTIONS:
Drug: WR 279,396 topical cream — WR 279,396 is a topical antibiotic cream containing 15% paromomycin and 0.5% gentamicin that will be applied to each lesion once a day and covered with a sterile gauze and tape dressing.
  Arms: WR 279,396 Topical Treament
Drug: Paromomycin Alone topical cream — The antibiotic paromomycin 15% in the same topical cream used in arm 1 will be applied to lesions daily and covered with a protective sterile gauze and tape dressing.
  Arms: Paromomycin Alone Topical treatment
Drug: Vehicle placebo cream — Applied daily to cutaneous leishmaniasis lesions, primarily ulcerative, and covered with a protective, sterile gauze and tape dressing.
  Arms: Vehicle Placebo Cream

SUMMARY:
This study will test the ability of the topical cream WR 279,396 to treat the skin lesions caused by the parasite called leishmania. WR 279,396 is an antibiotic preparation that contains paromomycin + gentamicin. This cream will be compared to the effect of a topical cream containing paromomycin alone and to a placebo cream that contains no antibiotics. Therefore, this study will have three groups of patients, and they will be assigned to one of these treatments randomly. The study will be carried out without the patient or the physician knowing which cream is being used for which patient. The goal is to determine if WR 279,396 cream or the paromomycin cream is better than placebo, and if WR 279,396 is better than paromomycin alone.

DETAILED DESCRIPTION:
This is an efficacy study to test the ability of WR 279,396 topical cream to treat uncomplicated cutaneous leishmaniasis caused primarily by Leishmania major in adults and children in Tunisia where the disease in endemic. A total of 375 volunteers will be randomized to the three arms described above to determine product efficacy. Safety data in all three arms will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* The subject was age 5 years or older, but less than 65 years.
* The subject was able to understand the information provided to him/her and give written informed consent. Consent was obtained from the parent/guardian of subjects who were < 18 years old. Children 12 to < 18 years old were asked to sign the written assent form. Witnessed verbal assent was obtained from subjects 5 to 11 years old.
* The subject was a male or female who was generally healthy.
* The subject had cutaneous lesions diagnosed as leishmaniasis in the index lesion by: (1) the identification of promastigotes in a culture of an aspirated lesion, or (2) the microscopic identification of Leishmania amastigotes on a DifQuik or Giemsa stained smear obtained from a lesion scraping.
* The subject had five or fewer cutaneous lesions.
* The subject had one lesion, which would be designated as the index lesion, that was ≥ 1 and < 5 cm in its greatest diameter and primarily ulcerative, ie, not purely verrucous or nodular.
* The subject was willing to forego other forms of treatment for CL, including other investigational treatment during the study.
* In the opinion of the principal investigator, the subject or subject's parent/guardian was capable of understanding and complying with the protocol

Exclusion Criteria

* The subject received previous treatment for leishmaniasis (including WR 279,396) within the last 6-months, with the exception of mercurochrome.
* The subject had difficulty complying with instructions on maintaining the dressing, eg, due to life style activities or age.
* The subject had only a single lesion whose characteristics included any of the following: verrucous or nodular lesion, ≥ 5 cm in its greatest diameter, < 1 cm or located on the ear, or other location that in the opinion of the principal investigator would be difficult to maintain application of study drug topically.
* The subject had a lesion due to Leishmania that involved the mucosa.
* The subject had signs or symptoms of disseminated disease, ie, clinically significant lymphadenitis with nodules that were painful and > 1 cm in the lymphatic drainage of the ulcer.
* The subject was a female with a positive urine pregnancy test, or who was breast feeding or lactating.
* The subject had an active malignancy or had a history of a solid, metastatic or hematologic malignancy, with the exception of a basal or squamous cell carcinoma of the skin that had been removed.
* The subject had a significant organ abnormality or chronic disease that, in the opinion of the investigator, would warrant exclusion of the subject from the study or would prevent the subject from completing the study.
* The subject was receiving any of the following medications: any medication containing pentavalent antimony, including stibogluconate sodium (Pentostam®) and meglumine antimoniate (Glucantime®); amphotericin B, including liposomal amphotericin B and amphotericin B deoxycholate; other medications containing paromomycin (administered IV or topically); methylbenzethonium chloride, fluconazole, ketoconazole, itraconazole; pentamidine; or allopurinol.
* The subject or the subject's parent/guardian was unable to understand verbal and/or written Arabic, English, or French (languages in which certified translations of the informed consent were available).
* The subject presented with an immuno-compromising condition, including recidivant leishmaniasis (during the past 2 years), or diabetes.
* The subject had a history of known or suspected idiosyncratic reactions or hypersensitivity to aminoglycosides.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2008-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afif Ben Salah, M.D., Ph.D., Principal Investigator — Institute Pasteur Tunisia
Locations (1):
- Central Clinic-Sidi Bouzid, Tunis, Tunisia

REFERENCES:
- [Derived] Ben Salah A, Ben Messaoud N, Guedri E, Zaatour A, Ben Alaya N, Bettaieb J, Gharbi A, Belhadj Hamida N, Boukthir A, Chlif S, Abdelhamid K, El Ahmadi Z, Louzir H, Mokni M, Morizot G, Buffet P, Smith PL, Kopydlowski KM, Kreishman-Deitrick M, Smith KS, Nielsen CJ, Ullman DR, Norwood JA, Thorne GD, McCarthy WF, Adams RC, Rice RM, Tang D, Berman J, Ransom J, Magill AJ, Grogl M. Topical paromomycin with or without gentamicin for cutaneous leishmaniasis. N Engl J Med. 2013 Feb 7;368(6):524-32. doi: 10.1056/NEJMoa1202657. PMID 23388004

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Started | 125 | 125 | 125
Completed | 123 | 122 | 103
Not Completed | 2 | 3 | 22
Not completed — Lost to Follow-up | 1 | 1 | 4
Not completed — Clinical failures | 1 | 0 | 12
Not completed — Withdrawal by investigator | 0 | 1 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream | Total
Number analyzed (Participants) | 125 | 125 | 125 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.4 (15.9) | 24.6 (15.7) | 23.2 (15.2) | 23.7 (15.6)
Age, Customized [Number; unit: participants]
  Adults | 63 | 66 | 61 | 190
  Children (12 to 17) | 24 | 33 | 35 | 92
  Children (5 to 11) | 38 | 26 | 29 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 57 | 56 | 182
  Male | 56 | 68 | 69 | 193
Race/Ethnicity, Customized [Number; unit: participants]
  North African | 125 | 125 | 125 | 375
Total Number of lesions per subject [Number; unit: participants]
  1 lesion | 59 | 49 | 50 | 158
  More than 1 lesions | 66 | 76 | 75 | 217
All lesion characteristics [Number; unit: lesions]
  Number of | 243 | 272 | 282 | 797
  Flat-like | 0 | 1 | 0 | 1
  Nodule | 0 | 1 | 0 | 1
  Other | 3 | 7 | 3 | 13
  Papule | 0 | 1 | 0 | 1
  Ulcerative | 240 | 262 | 279 | 781
Index lesion ulceration area [Mean (Standard Deviation); unit: mm^2] — Index lesion ulceration area per participant
  mm^2 | 126 (121) | 90.2 (74.5) | 97.7 (112) | 105 (105)
Index lesion [Number; unit: participants]
  Area of ulceration ≤ 100 m^2 | 72 | 84 | 89 | 245
  Area of ulceration > 100 mm^2 | 53 | 41 | 36 | 130
All lesion ulceration area [Mean (Standard Deviation); unit: mm^2] — Lesion ulceration area per lesion independent of participant
  mm^2 | 86.8 (107) | 65.6 (91.1) | 70.3 (91.4) | 73.8 (96.5)
All ulcerated lesions [Number; unit: lesions]
  Area of ulceration ≤ 100 m^2 | 175 | 210 | 222 | 607
  Area of ulceration > 100 mm^2 | 65 | 52 | 57 | 174
Days before treatment that index lesion was first noticed [Mean (Standard Deviation); unit: days] | 39.3 (25.7) | 39.5 (20.0) | 38.9 (20.5) | 39.2 (22.2)
Days before treatment that index lesion was first noticed (categorical) [Number; unit: participants]
  ≤ 60 days | 110 | 109 | 109 | 328
  > 60 days | 15 | 16 | 16 | 47

OUTCOME MEASURES:

1. Primary Outcome: Final Clinical Cure Rate
Description: Final clinical cure was defined as an index lesion that met the criteria for initial clinical cure without relapse. Definitions for index lesion outcomes were as follows:
  * Initial Clinical Improvement: At least 50% to 99% reduction in the size of the measured lesion from the baseline measurement by the Day 42 evaluation.
  * Initial Clinical Cure: 100% re-epithelialization (ie, a 0 x 0 length x width measurement) of the lesion at the nominal Day 42 evaluation, or initial clinical improvement followed by 100% re-epithelialization by Day 98.
  * Relapse: Initial clinical cure followed by re-ulceration by Day 168, or initial clinical improvement followed by lesion enlargement by Day 168.
  * Final Clinical Cure: Initial clinical cure without relapse through study Day 168.Clinical Failure: Lack of at least initial clinical improvement by Day 42, or relapse.
Time Frame: Day 42, 98, and 168
Population: Modified intention-to-treat (mITT) - all subjects randomized who received at least one treatment of study drug.
Measure: Number; unit: participants
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
participants | 101 | 102 | 73
Statistical Analysis 1: Comparison: WR 279,396 Topical Treament vs Vehicle Placebo Cream; H01: There is no difference in the final clinical cure rate between WR 279,396 and Vehicle AND there is no difference in the final clinical cure rate between Paromomycin Alone and Vehicle; Test type: Superiority or Other; p = 0.0001, Chi-squared
Statistical Analysis 2: Comparison: Paromomycin Alone Topical Treatment vs Vehicle Placebo Cream; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 3: Comparison: WR 279,396 Topical Treament vs Paromomycin Alone Topical Treatment; H02: There is no difference in clinical cure between WR 279,396 and Paromomycin Alone. Test of H02: If H01 was rejected, then H02 would be tested. The comparison of WR 279,396 versus Paromomycin Alone would be considered statistically significant if p < .05; Test type: Non-Inferiority or Equivalence — Test of H02: If H01 was rejected, then H02 would be tested. The comparison of WR 279,396 versus Paromomycin Alone would be considered statistically significant if p < .05; p = 0.871, Chi-squared

2. Secondary Outcome: Final Clinical Cure Rate (Per Protocol Dataset)
Description: Final clinical cure was defined as an index lesion that met the criteria for initial clinical cure without relapse. Definitions for index lesion outcomes as described in the primary outcome measure.
Time Frame: Day 42, 98, and 168
Population: Per protocol - all randomized subjects who received at least one treatment of study drug and whose outcomes at Day 42, Day 98 (if applicable) and Day 168 could be assessed. However, a subject was still considered per-protocol if withdrawn early for treatment failure.
Measure: Number; unit: participants
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 124 | 120
participants | 101 | 102 | 73
Statistical Analysis 1: Comparison: WR 279,396 Topical Treament vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.0006, Chi-squared
Statistical Analysis 2: Comparison: Paromomycin Alone Topical Treatment vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.0002, Chi-squared
Statistical Analysis 3: Comparison: WR 279,396 Topical Treament vs Paromomycin Alone Topical Treatment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.767, Chi-squared

3. Secondary Outcome: Estimated Percentage Subjects With Re-epithelialization of the Index Lesion Without Relapse
Description: For the first of the above analyses, subjects were considered to have endpoint events at the first assessment on or before Day 42 where complete re-epithelialization occurred at the index lesion that was not followed by a later assessment where ulceration was present. Subjects who did not have complete re-epithelialization by Day 42 or who relapsed after Day 42 were censored in the analysis at the Day 42 assessment. This analysis was only to be conducted through Day 42.
Time Frame: Day 42
Population: mITT dataset
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
percentage of participants | 67.2 [58.5 to 74.8] | 68.8 [60.2 to 76.3] | 48.8 [40.2 to 57.5]
Statistical Analysis 1: Comparison: WR 279,396 Topical Treament vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.330, Log Rank; Mantel-Cox (log-rank) grouped failure time test using proportion re-epithelialized at each of the scheduled assessments through Day 42 without relapse
Statistical Analysis 2: Comparison: Paromomycin Alone Topical Treatment vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.275, Log Rank
Statistical Analysis 3: Comparison: WR 279,396 Topical Treament vs Paromomycin Alone Topical Treatment; Test type: Non-Inferiority or Equivalence — The comparison of WR 279,396 versus Paromomycin Alone would be considered statistically significant if p < .05; p = 0.830, Log Rank

4. Secondary Outcome: Estimated Percentage of Subjects With Re-epithelialization of the Index Lesion Without Relapse at Various Times of Follow-up
Time Frame: Days 42, 49, and 98
Population: mITT dataset. The data show that 95.8% of the Vehicle-treated subjects remaining in the study at Day 168 (the percentage excludes the 17.6% of subjects who dropped out or were withdrawn early due to treatment failure) had re-epithelialization of the index lesion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
percentage of participants
  Day 42 | 67.2 [59.5 to 76.0] | 68.5 [60.8 to 77.2] | 49.4 [41.1 to 59.3]
  Day 49 | 72.9 [65.5 to 81.2] | 81.5 [74.9 to 88.6] | 57.1 [48.7 to 67.0]
  Day 98 | 94.3 [90.3 to 98.5] | 99.2 [97.6 to 100.0] | 90.9 [85.3 to 96.8]

5. Secondary Outcome: Estimated Percentage of All Treated Ulcerated Lesions Without Relapse at Day 42
Time Frame: Days 42
Population: mITT dataset
Measure: Number (95% Confidence Interval); unit: Percentage of lesions
Units Other Than Participants: lesions
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
Number analyzed (lesions) | 157 | 134 | 115
Percentage of lesions | 51.7 [45.7 to 58.4] | 81.6 [77.0 to 86.4] | 58.1 [52.4 to 64.4]

6. Secondary Outcome: Estimated Percentage of All Treated Ulcerated Lesions Without Relapse at Day 49
Time Frame: Days 49
Population: mITT dataset
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
Number analyzed (lesions) | 56 | 42 | 67
percentage of lesions | 81.4 [76.6 to 86.5] | 90.4 [86.9 to 94.1] | 64.9 [59.2 to 71.1]

7. Secondary Outcome: Estimated Percentage of All Treated Ulcerated Lesions Without Relapse at Day 98
Time Frame: Days 98
Population: mITT dataset
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
Number analyzed (lesions) | 23 | 10 | 36
percentage of lesions | 91.5 [88.1 to 95.1] | 98.9 [97.6 to 100.0] | 92.2 [88.6 to 96.0]

8. Secondary Outcome: Number of Subjects Achieving Initial Clinical Improvement of the Index Lesion
Time Frame: Day 42
Measure: Number; unit: participants
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
participants | 105 | 107 | 77
Statistical Analysis 1: Comparison: WR 279,396 Topical Treament vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.0001, Chi-squared
Statistical Analysis 2: Comparison: Paromomycin Alone Topical Treatment vs Vehicle Placebo Cream; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 3: Comparison: WR 279,396 Topical Treament vs Paromomycin Alone Topical Treatment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.725, Chi-squared

9. Secondary Outcome: Number of Subjects Achieving Re-epithelialization of the Index Lesion Without Relapse
Description: Number of Subjects Achieving Re-epithelialization of the Index Lesion by Day 42 without Relapse from Day 42 Onward, Imputing Relapse for any Subject with a Missing Visit after Day 42
Time Frame: Day 168
Population: mITT population
Measure: Number; unit: participants
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
participants | 84 | 84 | 62
Statistical Analysis 1: Comparison: WR 279,396 Topical Treament vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.005, Chi-squared
Statistical Analysis 2: Comparison: Paromomycin Alone Topical Treatment vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.005, Chi-squared
Statistical Analysis 3: Comparison: WR 279,396 Topical Treament vs Paromomycin Alone Topical Treatment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p = 1.000, Chi-squared

10. Secondary Outcome: Number of Subjects Achieving Re-epithelialization of All Treated Ulcerated Lesions Without Subsequent Relapse
Description: Number of Subjects Achieving Re-epithelialization of All Treated Ulcerated Lesions at Day 42 without Subsequent Relapse from Day 42 Onward,
Time Frame: Day 168
Population: mITT dataset
Measure: Number; unit: participants
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
participants | 83 | 84 | 60
Statistical Analysis 1: Comparison: WR 279,396 Topical Treament vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.003, Chi-squared
Statistical Analysis 2: Comparison: Paromomycin Alone Topical Treatment vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.002, Chi-squared
Statistical Analysis 3: Comparison: WR 279,396 Topical Treament vs Paromomycin Alone Topical Treatment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.893, Chi-squared

11. Secondary Outcome: Number of All Ulcerated Lesions Achieving 100% Re-epithelialization by Day 42
Time Frame: Day 42
Population: mITT dataset
Measure: Number; unit: Ulcerated lesions
Units Other Than Participants: Ulcerated lesions
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
Number analyzed (Ulcerated lesions) | 240 | 262 | 279
Ulcerated lesions | 190 | 218 | 160
Statistical Analysis 1: Comparison: WR 279,396 Topical Treament vs Vehicle Placebo Cream; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Paromomycin Alone Topical Treatment vs Vehicle Placebo Cream; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: WR 279,396 Topical Treament vs Paromomycin Alone Topical Treatment; Test type: Non-Inferiority or Equivalence — The comparison of WR 279,396 versus Paromomycin Alone would be considered statistically significant if p < .05; p = 0.247, Chi-squared

12. Secondary Outcome: Number of Subjects With a Relapse on or After Day 42
Time Frame: Day 168
Measure: Number; unit: participants
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Number analyzed (Participants) | 125 | 125 | 125
participants | 4 | 3 | 2
Statistical Analysis 1: Comparison: WR 279,396 Topical Treament vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.409, Chi-squared
Statistical Analysis 2: Comparison: Paromomycin Alone Topical Treatment vs Vehicle Placebo Cream; Test type: Superiority or Other; p = 0.651, Chi-squared
Statistical Analysis 3: Comparison: WR 279,396 Topical Treament; Test type: Non-Inferiority or Equivalence — The comparison of WR 279,396 versus Paromomycin Alone would be considered statistically significant if p < .05; p = 0.701, Chi-squared

ADVERSE EVENTS:
Time Frame: 168 day follow up
Arm/Group | WR 279,396 Topical Treament | Paromomycin Alone Topical Treatment | Vehicle Placebo Cream
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/125 | 0/125
Other Adverse Events (participants affected / at risk) | 55/125 | 51/125 | 45/125
OTHER ADVERSE EVENTS (reported when occurring in more than 0.8% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | WR 279,396 Topical Treament (N=125) | Paromomycin Alone Topical Treatment (N=125) | Vehicle Placebo Cream (N=125)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Application site bleeding (General disorders) | 1 | 0 | 0
Application site erythema (General disorders) | 6 | 7 | 4
Application site infection (Gastrointestinal disorders) | 1 | 0 | 2
Application site pain (General disorders) | 1 | 1 | 0
Application site vesicles (General disorders) | 31 | 32 | 9
Oedema (General disorders) | 2 | 3 | 5
Pain (General disorders) | 2 | 2 | 1
Bronchitis (Infections and infestations) | 5 | 3 | 5
Paronychia (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0
Superinfection (Infections and infestations) | 3 | 0 | 12
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Headache (Nervous system disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 5 | 9 | 6
Vein pain (Vascular disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Breast abscess (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1
Mumps (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Application site inflammation (Infections and infestations) | 0 | 0 | 2
Cellulitis (Immune system disorders) | 0 | 0 | 1
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No